CLINICAL TRIAL: NCT05403255
Title: Quality of Life and Psychosocial Dimensions in Children With Congenital or Acquired Hypopituitarism
Brief Title: Quality of Life and Psychosocial Dimension in Children With Hypopituitarism
Acronym: QALHYPO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00504-39
Record Dates: First submitted 2022-05-17; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Congenital or Acquired Hypopituitarism
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple or isolated pituitary hormone deficiency group: Patient with multiple pituitary deficiency or isolated pituitary deficiency diagnosed for at least 6 months.
  Interventions: Other: evaluation of the quality of life with questionnaires

INTERVENTIONS:
Other: evaluation of the quality of life with questionnaires — Questionnaire data will be collected among patients and their parents during follow-up consultations.
  Children's quality of life will be evaluated using the Kidscreen-10 questionnaire (for children and parents) and PedsQL multidimensional fatigue scale. Psychosocial indicators (standard of living, schooling, recreation activities, social and family relationships, perceived health status and physical appearance) will be gathered using a questionnaire based on the HBSC (Health Behaviour in School-Aged Children) questionnaire (INPES 2010), and compared with data from the general population of elementary-, middle-and high-school children in France.

SUMMARY:
Relatively little is known about the quality of life (QOL) of patients with hypopituitarism, particularly children. Quality of life studies have mostly focused on improvements following the initiation of growth hormone treatment in adults with growth hormone deficiency. Overall QOL data on patients with multiple pituitary hormone deficiency or another isolated deficiency are much scarcer. These studies suggest however that pituitary deficiencies affect the QOL and social integration of adults. In children, the psychosocial repercussions of the disease are very poorly understood, particularly in the case of multiple congenital pituitary hormone deficiency.

DETAILED DESCRIPTION:
Objectives:

* Describe the quality of life and psychosocial repercussions of the disease in children 10-17 years of age with multiple pituitary hormone deficiency (either acquired or congenital), or isolated pituitary hormone deficiency (other than idiopathic isolated growth hormone deficiency).
* Compare the QOL and psychosocial indicators of these patients with those of the general population
* Study the effects of various factors (medical, social, psychological) on patient outcomes and experiences of the disease.

Methods

* Prospective analytical pilot study involving the four hospitals in the Referral Centre for Rare Pituitary Diseases (Centre de Référence des Maladies Rares de l'Hypophyse, HYPO)
* Questionnaire data will be collected among patients and their parents during follow-up consultations.
* Children's quality of life will be evaluated using the Kidscreen-10 questionnaire (for children and parents) and PedsQL multidimensional fatigue scale. Psychosocial indicators (standard of living, schooling, recreation activities, social and family relationships, perceived health status and physical appearance) will be gathered using a questionnaire based on the HBSC (Health Behaviour in School-Aged Children) questionnaire (INPES 2010), and compared with data from the general population of elementary-, middle-and high-school children in France.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 years
* Multiple or isolated pituitary hormone deficiency
* Deficiency diagnosed for a least 6 months

Exclusion Criteria:

* Isolated growth hormone deficiency with normal MRI findings and/or no previous irradiation of the hypothalamo-pituitary region and/or no known genetic cause.
* Secondary pituitary deficiency due to a secreting adenoma
* Inability to complete the questionnaire (intellectual disability, low French language proficiency)
* No health coverage

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The research involves the inclusion of special populations. Indeed, the research plans to include 120 patients aged 10 to 17 years.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life measurement | 1 day
  The KIDSCREEN-10 score consists of 10 items and provides a Rasch-scaled single score of HRQoL. Both self-report and proxy versions will be used.

SECONDARY OUTCOMES:
Psychosocial parameters | 1 day
  HBSC questionnaires (Aged Behaviour in School-agedd Children, INPES 2014). This international standard questionnaire enables the collection of common data across participating countries and thus enables the quantification of patterns of key health behaviours, health indicators and contextual variables.
Socioeconomic status | 1 day
  ENVU questionaire ( Social and health vulnerability identification questionnaire in pediatrics )
Fatigue | 1 day
  PedsQL multidimensional fatigue scale

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — ASSISTANCE PUBLIQUE HOPITAUX MARSEILLE; Sarah CASTETS, PH, Principal Investigator — ASSISTANCE PUBLIQUE HOPITAUX MARSEILLE
Locations (1):
- Assistance Publique Hopitaux Marseille, Marseille, Bouches-du-Rhône, France